CLINICAL TRIAL: NCT03047603
Title: Evaluation of Diagnostic and Differential Diagnostic Significance of a Combination of PIVKA-II and Other Tumor Markers in Hepatocellular Carcinoma
Brief Title: Evaluation of Diagnostic Efficiency of PIVKA-II and Other Tumor Markers in HCC
Status: Completed | Type: Observational
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Collaborators: Abbott Diagnostics Division (Industry); Peking University First Hospital (Other); The First Hospital of Jilin University (Other); RenJi Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Gansu Provincial Hospital (Other); Henan Provincial People's Hospital (Other); Sun Yat-sen University (Other); Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Tian Yang, Doctor,Associate professor, Eastern Hepatobiliary Surgery Hospital
Other Study IDs: Pivkaii
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Protein induced by vitamin K absence or antagonist-II; Differential diagnosis; Des-γ-carboxy prothrombin; Alpha-fetoprotein; Lens culinaris agglutinin-reactive fraction of alpha-fetoprotein-fetoprotein
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy control: The healthy control group consist of people undergoing routine medical examination. Serum samples are collected.
  Interventions: Diagnostic Test: PIVKA-II
- Metastatic liver cancer patients: Serum samples are collected.
  Interventions: Diagnostic Test: PIVKA-II
- Hepatocellular carcinoma patients: Serum samples are collected before liver resection.
  Interventions: Diagnostic Test: PIVKA-II
- Chronic liver disease patients: This group is comprised of liver cirrhosis and chronic hepatitis B patients. The diagnosis of liver cirrhosis are based on triple-phase contrast enhanced computed tomography, magnetic resonance imaging.
  Interventions: Diagnostic Test: PIVKA-II

INTERVENTIONS:
Diagnostic Test: PIVKA-II — Serum samples are tested for tumor markers including PIVKA-II,AFP,AFP-L3% and biochemical tests.
  Other Names: DCP

SUMMARY:
The incidence of Hepatocellular carcinoma (HCC) is increasing worldwide. However, most of HCC cases were at advanced stage when the diagnosis established.Early diagnosis improves the prognosis.The study is intended to evaluate the diagnostic efficiency of Protein Induced by Vitamin K Absence or antagonist-II(PIVKA-II). This study is a international multicenter study joined by several hospitals in China,Singapore,Thailand and Vietnam. Participants including healthy control,HCC,metastatic liver cancer,Hepatitis B virus(HBV) and liver cirrhosis are consecutively recruited into the cohort. All the serum samples are collected before any treatments and will be tested in single center in order to decrease bias. Serum samples were tested for PIVKA-II,alpha-fetoprotein and biochemical indexes including alanine aminotransferase(ALT),aspartate aminotransferase(AST),gamma-glutamyl transferase(GGT),alpha-l-fucosidase(AFU),etc.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third leading cause of cancer deaths worldwide.Early diagnosis improves the prognosis. Protein induced by vitamin K antagonist-II (PIVKA-II), also known as des-γ-carboxyprothrombin (DCP) or acarboxy prothrombin, is an abnormal form of prothrombin induced by vitamin K absence or antagonist-II. The study is intended to evaluate the diagnostic efficiency of Protein Induced by Vitamin K Absence or antagonist-II(PIVKA-II). PIVKA-II as an effective tumor marker for hepatocellular carcinoma(HCC) has been widely used in the western countries where most cases are hepatitis C virus(HCV) related.However, the majority of HCCs in China are HBV related. Despite the extensive application of PIVKA-II in some hospitals from China, the diagnostic efficiency including sensitivity,specificity,positive predictive value and negative predictive value still needs more clinical data to evaluate. The research purposes list as follows：1.Determination of diagnostic Cut-off value 2.Evaluation of diagnostic efficiency of PIVKA-II 3.Evaluation of the combination of PIVKA-II and other tumor markers for HCC. This study is an international multicenter study joined by several hospitals in China,Singapore,Thailand and Vietnam. Participants including healthy control,HCC,metastatic liver cancer,HBV and liver cirrhosis are consecutively recruited into the cohort. All the serum samples are collected before any treatments and will be tested in single center in order to decrease bias. Serum samples were tested for PIVKA-II,Alpha-fetoprotein(AFP)，alpha-fetoprotein L3 and biochemical indexes including ALT,AST,GGT,AFU,etc. The diagnosis of HCC was based on histopathology. All HCC diagnoses were confirmed at the time of analysis.The Student's t-test (or Mann-Whitney test) was used to compare continuous variables, and the chi-square test (or Fisher's exact test) was used for categorical variables. A receiver operator characteristic (ROC) curve was used to assess the performance characteristic of PIVKA-II,AFP,AFP-L3 measurement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85
* Receiving no treatment before diagnosis
* Establishing Diagnosis according to the Asian Pacific Association for the Study of Liver(APASL) criteria

Exclusion Criteria:

* Clinical data missing
* Laboratory tests information missing
* Serum samples doesn't qualified
* Obstructive jaundice patients
* Medical history of taking warfarin

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited through outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 4005 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
PIVKA-II | Day one
  Using PIVKA-II assay kit(chemiluminescent microparticle immunoassay).

SECONDARY OUTCOMES:
AFP,AFP-L3% | Day one
ALT, AST，γ-GT， AFU | Day one

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobiliary surgery hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yang T, Xing H, Wang G, Wang N, Liu M, Yan C, Li H, Wei L, Li S, Fan Z, Shi M, Chen W, Cai S, Pawlik TM, Soh A, Beshiri A, Lau WY, Wu M, Zheng Y, Shen F. A Novel Online Calculator Based on Serum Biomarkers to Detect Hepatocellular Carcinoma among Patients with Hepatitis B. Clin Chem. 2019 Dec;65(12):1543-1553. doi: 10.1373/clinchem.2019.308965. Epub 2019 Oct 31. PMID 31672853
- [Derived] Yan C, Hu J, Yang J, Chen Z, Li H, Wei L, Zhang W, Xing H, Sang G, Wang X, Han R, Liu P, Li Z, Li Z, Huang Y, Jiang L, Li S, Dai S, Wang N, Yang Y, Ma L, Soh A, Beshiri A, Shen F, Yang T, Fan Z, Zheng Y, Chen W. Serum ARCHITECT PIVKA-II reference interval in healthy Chinese adults: Sub-analysis from a prospective multicenter study. Clin Biochem. 2018 Apr;54:32-36. doi: 10.1016/j.clinbiochem.2018.02.007. Epub 2018 Feb 12. PMID 29448045
- [Derived] Yan C, Yang J, Wei L, Hu J, Song J, Wang X, Han R, Huang Y, Zhang W, Soh A, Beshiri A, Fan Z, Zheng Y, Chen W. Serum reference interval of ARCHITECT alpha-fetoprotein in healthy Chinese Han adults: Sub-analysis of a prospective multi-center study. Clin Biochem. 2018 Feb;52:164-166. doi: 10.1016/j.clinbiochem.2017.11.002. Epub 2017 Nov 10. PMID 29129627